CLINICAL TRIAL: NCT02581943
Title: Immune Response in Patients With Recurrent or Metastatic Non-small Cell Lung Cancer and Performance Status of 2 Treated With a Combination of Pembrolizumab and Low Dose Weekly Carboplatin/Paclitaxel
Brief Title: Effect of Pembrolizumab With or Without Carboplatin and Paclitaxel on Immune Response in Patients With Recurrent or Stage IIIB-IV Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00034830; NCI-2015-01708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU #62415; CCCWFU 62415 (Other: Wake Forest University Health Sciences); P30CA012197 (NIH)
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-12

CONDITIONS: Recurrent Non-Small Cell Lung Carcinoma; Stage IIIB Non-Small Cell Lung Cancer; Stage IV Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Paclitaxel; Taxes; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab; Other: Quality-of-Life Assessment
- Arm II (pembrolizumab, paclitaxel, carboplatin) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1, paclitaxel IV over 1 hour and carboplatin IV over 1 hour on days 1, 7 and 14. Courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carboplatin; Other: Laboratory Biomarker Analysis; Drug: Paclitaxel; Biological: Pembrolizumab; Other: Quality-of-Life Assessment

INTERVENTIONS:
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplat; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
  Arms: Arm II (pembrolizumab, paclitaxel, carboplatin)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
  Arms: Arm II (pembrolizumab, paclitaxel, carboplatin)
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment

SUMMARY:
This randomized pilot phase II trial studies the effect of pembrolizumab with or without carboplatin and paclitaxel on immune response in patients with non-small cell lung cancer that has come back or stage IIIB-IV. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as carboplatin and paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving pembrolizumab together with carboplatin and paclitaxel may improve immune responses in patients with non-small cell lung cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the immune effects of single agent pembrolizumab and pembrolizumab combined with low-dose carboplatin and paclitaxel.

II. Estimate the treatment response to single agent pembrolizumab and pembrolizumab combined with low-dose carboplatin and paclitaxel.

SECONDARY OBJECTIVES:

I. Determine the toxicity and tolerability of pembrolizumab and pembrolizumab combined with low-dose carboplatin and paclitaxel.

II. Assess quality of life (QOL) in patients receiving single agent pembrolizumab and pembrolizumab combined with carboplatin and paclitaxel.

III. Assess the association between immune response and clinical response.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1.

ARM II: Patients receive pembrolizumab IV over 30 minutes on day 1, paclitaxel IV over 1 hour and carboplatin IV over 1 hour on days 1, 7 and 14.

In both arms, courses repeat every 3 weeks for 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for at least 30 days and then every 8 weeks thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed non-small cell lung cancer (NSCLC) that is advanced/metastatic (stage IIIB/IV) or recurrent (progression after surgery or radiation or chemo-radiation treatment for loco-regional disease). Patients with epidermal growth factor (EGFR) mutation, anaplastic lymphoma kinase (ALK) gene rearrangement or ROS1 translocation must have received an approved EGFR, ALK, or ROS1-directed therapy and have signs of disease progression prior to receiving pembrolizumab.
* Patients must be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion; newly-obtained is defined as a specimen obtained up to 12 weeks (84 days) prior to date of signing consent.
* Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen (up to 3 years) only upon agreement from the Sponsor. At least 4 mm of tumor tissue will be needed for PD-L1 staining.
* Patients who have received zero (0) to two (2) previous lines of systemic chemotherapy and are not currently receiving chemotherapy treatment (within 2 weeks of randomization).
* At least one measurable lesion as defined by RECIST v1.1 on screening computed tomography (CT) or magnetic resonance imaging (MRI)
* Age >18 years.
* ECOG performance status of 2.
* Patients must have normal organ and marrow function as defined below:
* white blood cell count > 2,500 cells/mcL
* absolute neutrophil count >1,500/mcL
* platelets >100,000/mcL
* hemoglobin ≥ 9 g/dL
* total bilirubin ≤ 2.0 x upper limit of normal (ULN)
* AST(SGOT)/ALT(SGPT) < 2.5 x ULN Or ≤ 5 x ULN in presence of liver metastases
* creatinine within normal institutional limits OR
* creatinine clearance > 50 mL/min for patients with creatinine levels above institutional normal
* potassium ≥ lower limit of normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for the duration of study participation and for 4 weeks after the final administration of study drugs. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign an IRB-approved informed consent document.

Exclusion Criteria

* Known active (untreated) central nervous system (CNS) metastases that require steroids. Subjects with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for at least 2 weeks before study entry, defined as:

  * No evidence of new or enlarging CNS metastasis or new neurological symptoms attributable to CNS metastases.
  * Asymptomatic and receiving either no or stable doses of anticonvulsants and total doses of corticosteroids equivalent to 10 mg of prednisone or less.
* Current or previous other malignancy within 2 years of study entry, except cured basal or squamous cell skin cancer, superficial bladder cancer, prostate intraepithelial neoplasm, carcinoma in situ of the cervix, or other noninvasive or indolent malignancy without sponsor approval.
* History of previous exposure to an anti PD1/PD-L1 agent
* Patients receiving any other investigational agents and or more than two different chemotherapy regimens for treatment of metastatic disease.
* Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.
* Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
* Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab, paclitaxel or carboplatin.
* Current uncontrolled cardiac disease such as angina or myocardial infarction, congestive heart failure including New York Heart Association functional classification of 3, or arrhythmia requiring treatment.
* History of pneumonitis or active lung infection.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungals, or antivirals.
* Patients receiving chronic steroids and or immunosuppression.
* Known HIV infection, Hepatitis B virus (HBV) or hepatitis C virus (HCV) viremia or at risk for HBV reactivation. HBV DNA and testing for HCV RNA must be undetectable. At risk for HBV reactivation is defined as hepatitis B surface antigen positive or anti-hepatitis B core antibody positive.
* History of autoimmune disease(s).
* Psychiatric illness/social situations that would limit compliance with study requirements.
* Any other condition or circumstance that could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives such as history of, or any evidence of active, non-infectious pneumonitis.
* Has an active infection requiring systemic therapy.
* Pregnant women are excluded from this study because of the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants, breastfeeding should be discontinued prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2022-11-19 (Actual); Study Completion 2022-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William J Petty, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Started | 22 | 21
Completed | 4 | 2
Not Completed | 18 | 19
Not completed — Death | 5 | 2
Not completed — Disease Progression | 12 | 15
Not completed — Withdrawal by Subject | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin) | Total
Number analyzed (Participants) | 22 | 21 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.5 (8.7) | 70.8 (11.1) | 70.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 12 | 19
  Male | 15 | 9 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 19 | 18 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Duration of Response
Description: Duration of response will also be assessed in each group and compared using survival analysis methods. Per response evaluation criteria in Solid Tumors Criteria: Complete Response (irCR): Complete disappearance of all target and new, measurable lesions, with the exceptions of lymph nodes which must decrease to < 10 mm in short axis; Partial Response (irPR): Decrease in TMTB ≥ 30% relative to baseline; Stable Disease (irSD): Not meeting criteria for irCR or irPR, in absence of irPD; Progressive Disease (irPD): Increase in TMTB ≥ 20% relative to nadir.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 22 | 21
days | 98 [0 to 326] | 69 [0 to 252]
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Other; p = 0.366, Log Rank

2. Primary Outcome: Change in Effect of Treatment in Immune Markers From Baseline to End of Treatment (up to 2 Years)
Description: Immune markers were measured at baseline and post-treatment. Data reported are the difference (post-pre) in these immune markers. Wilcoxon rank-sum tests were used to analyze the effects of the treatments on the change in immune markers.
Time Frame: Baseline and end of treatment (up to 2 years)
Measure: Median (Inter-Quartile Range); unit: cells
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 10 | 9
cells
  CD4+FoxP3 | 1.82 [-2.11 to 4.73] | -1.34 [-3.37 to 269]
  MDSC | -3.83 [-6.47 to 0.92] | 5.41 [1.64 to 9.65]
  CD4+ICOS | 1.07 [0.02 to 2.10] | 5.41 [-0.64 to 5.70]
  CD8+ICOS | 0.7 [0.01 to 0.97] | 0.77 [-0.02 to 2.91]
  Plamacytoid DC | -0.17 [-1.85 to 0.04] | -0.02 [-0.38 to 0.19]
  Monocytes | -2.05 [-8.40 to -0.08] | 0.65 [-0.98 to 3.40]
  T cells (CD3+) | -13.06 [-25.72 to 22.62] | -0.01 [-16.60 to 12.16]
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.327, Wilcoxon (Mann-Whitney); test for CD4+FoxP3
Statistical Analysis 2: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.142, Wilcoxon (Mann-Whitney); test for MDSC
Statistical Analysis 3: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.462, Wilcoxon (Mann-Whitney) — test for CD4+ICOS+
Statistical Analysis 4: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.870, Wilcoxon (Mann-Whitney) — test for CD8+ICOS+
Statistical Analysis 5: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.414, Wilcoxon (Mann-Whitney) — test for Plamacytoid DC
Statistical Analysis 6: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.121, Wilcoxon (Mann-Whitney) — test for Monocytes
Statistical Analysis 7: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Equivalence — Null hypothesis: no difference between treatment arms in the post-pre difference in cell counts; p = 0.624, Wilcoxon (Mann-Whitney) — test for T cells (CD3+)

3. Primary Outcome: Objective Response Rate (ORR), Assessed Using RECIST
Description: The Fisher's exact test methods will be used to estimate ORR between groups. The Exact Clopper-Pearson 95% confidence intervals will be calculated for each group. Per response evaluation criteria in Solid Tumors Criteria: Complete Response (irCR): Complete disappearance of all target and new, measurable lesions, with the exceptions of lymph nodes which must decrease to < 10 mm in short axis; Partial Response (irPR): Decrease in TMTB ≥ 30% relative to baseline; Stable Disease (irSD): Not meeting criteria for irCR or irPR, in absence of irPD; Progressive Disease (irPD): Increase in TMTB ≥ 20% relative to nadir.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 22 | 21
Participants | 6 | 9
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Other; p = 0.348, Fisher Exact

4. Primary Outcome: Overall Survival
Description: The Kaplan Meier curves will be used to estimate overall survival rates.
Time Frame: Duration of time from randomization to the time of death due to any cause, or the date the subject was last confirmed to be alive, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 22 | 21
months | 8.4 [5.0 to 29.8] | 7.5 [3.9 to 25.1]
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Other; p = 0.63, Log Rank

5. Primary Outcome: Progression Free Survival
Description: The Kaplan Meier curves will be used to estimate progression free survival rates. Per response evaluation criteria in Solid Tumors Criteria: Progressive Disease (irPD): Increase in TMTB ≥ 20% relative to nadir.
Time Frame: Duration of time from randomization to the time of immune-related progressive disease or death, whichever comes first, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 22 | 21
months | 4.3 [1.9 to 12.0] | 5.0 [1.9 to 10.4]
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Other; p = 0.692, Log Rank

6. Secondary Outcome: Number of Participants With Reported Adverse Events - CTCAE Version 4.0
Description: Adverse events will be categorized by organ system and severity and summarized as frequency counts and percentages. A treatment will be considered too toxic if ≥6 of 20 patients in a cohort are removed from study because of toxicity.
Time Frame: At baseline, at week 8, week 12, week 20 and up to 30 days after last study drug is administered
Measure: Number; unit: participants with adverse event
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
Number analyzed (Participants) | 22 | 21
participants with adverse event | 21 | 18
Statistical Analysis 1: Comparison: Arm I (Pembrolizumab) vs Arm II (Pembrolizumab, Paclitaxel, Carboplatin); Test type: Other; p = 0.345, Fisher Exact

7. Secondary Outcome: Change in Immune Markers From Baseline to End of Treatment (up to 2 Years) With Treatment Response
Description: Treatment response will be grouped into 3 categories as defined earlier in the protocol (complete or partial response, stable disease, progressive disease). The immune responses for patients within each of these 3 groups will be examined to determine whether there is evidence of an association. Immune markers were measured at baseline and post-treatment. Data reported are the difference (post-pre) in these immune markers. The change in markers (post-pre) are summarized and compared between treatment groups using a Kruskal Wallis test.
Time Frame: At baseline and post-treatment
Measure: Median (Inter-Quartile Range); unit: Cells
Groups:
- Complete or Partial Response: Best response to treatment was complete or partial response
- Stable Disease: Best response to treatment was stable disease
- Progressive Disease: Disease progression with no response to treatment.
Arm/Group | Complete or Partial Response | Stable Disease | Progressive Disease
Number analyzed (Participants) | 9 | 4 | 5
Cells
  CD4+FoxP3 | -0.54 [-2.8 to 3.7] | -1.4 [-2.8 to 1.7] | -2.1 [-5.1 to 4.2]
  MDSC | 5.3 [-6.5 to 9.7] | -1.5 [-7.6 to 3.5] | -0.9 [-4.1 to 0.9]
  CD4+ICOS | 2.1 [1.2 to 5.6] | 3.2 [0.5 to 11.0] | 0.02 [-1.9 to 0.8]
  CD8+ICOS | 1.0 [0.01 to 3.5] | 1.9 [-0.9 to 6.4] | -0.02 [-0.3 to 0.1]
  Plamacytoid DC | -0.24 [-1.03 to 0.04] | 0.20 [-0.91 to 4.38] | -0.22 [-0.38 to -0.12]
  Monocytes | 0.65 [-2.71 to 3.40] | -0.36 [-4.50 to 6.17] | -1.75 [-11.47 to -0.08]
  T cells (CD3+) | -16.6 [-23.6 to -2.5] | 8.3 [2.2 to 17.4] | 1.4 [-23.9 to 32.0]
Statistical Analysis 1: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.917, Kruskal-Wallis; Test for CD8+ICOS
Statistical Analysis 2: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.746, Kruskal-Wallis; test for MDSC
Statistical Analysis 3: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.302, Kruskal-Wallis — test for CD4+ICOS
Statistical Analysis 4: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.130, Kruskal-Wallis; test for CD8+ICOS+
Statistical Analysis 5: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.628, Kruskal-Wallis — test for Plamacytoid DC
Statistical Analysis 6: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.567, Kruskal-Wallis — test for Monocytes
Statistical Analysis 7: Comparison: Complete or Partial Response vs Stable Disease vs Progressive Disease; Test type: Other; p = 0.311, Kruskal-Wallis — test for T cells (CD3+)

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm I (Pembrolizumab) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin)
All-Cause Mortality (participants affected / at risk) | 18/22 | 18/21
Serious Adverse Events (participants affected / at risk) | 3/22 | 3/21
Other Adverse Events (participants affected / at risk) | 21/22 | 18/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pembrolizumab) (N=22) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin) (N=21)
Death (General disorders) | 3 (3) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Pembrolizumab) (N=22) | Arm II (Pembrolizumab, Paclitaxel, Carboplatin) (N=21)
WBC decreased (Blood and lymphatic system disorders) | 10 (109) | 10 (129)
Platelets decreased (Blood and lymphatic system disorders) | 10 (111) | 10 (129)
Anemia (Blood and lymphatic system disorders) | 11 (112) | 11 (130)
Nausea (Gastrointestinal disorders) | 5 (13) | 8 (47)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 3 (6) | 6 (9)
Anorexia (Metabolism and nutrition disorders) | 4 (9) | 5 (9)
Alkaline phosphatase increased (Investigations) | 10 (110) | 11 (130)
Creatinine increased (Investigations) | 2 (2) | 1 (2)
Hypotension (Vascular disorders) | 3 (4) | 1 (2)
Neutrophil count decreased (Investigations) | 10 (108) | 10 (129)
Pain at administration site (General disorders) | 8 (44) | 8 (46)
Insomnia (Psychiatric disorders) | 3 (6) | 4 (22)
Fatigue (General disorders) | 12 (51) | 10 (58)
Hyperglycemia (Metabolism and nutrition disorders) | 10 (39) | 12 (66)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5) | 8 (25)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 4 (7) | 7 (20)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2) | 7 (17)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (22) | 13 (63)
Bilirubin increased (Investigations) | 10 (50) | 10 (55)
Alanine aminotranspherase increased (Investigations) | 10 (53) | 11 (56)
Constipation (Gastrointestinal disorders) | 3 (10) | 5 (9)
Aspartate aminotranspherase increased (Investigations) | 10 (54) | 11 (56)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (12) | 6 (17)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Confusion (Psychiatric disorders) | 2 (3) | 2 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 1 (1) | 4 (8)
Lymphocyte count decreased (Investigations) | 4 (6) | 6 (29)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Blurred Vision (Eye disorders) | 2 (2) | 1 (1)
Edema limbs (General disorders) | 2 (7) | 7 (26)
Abdominal Pain (Gastrointestinal disorders) | 3 (4) | 0 (0)
Mucositis Oral (Gastrointestinal disorders) | 1 (4) | 0 (0)
Non-cardiac chest pain (General disorders) | 5 (12) | 1 (2)
Sinusitis (Infections and infestations) | 2 (3) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 3 (3)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 4 (8) | 4 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 2 (2) | 7 (12)
Peripheral Sensory Neuropathy (Nervous system disorders) | 1 (1) | 3 (9)
Acute Kidney Injury (Renal and urinary disorders) | 3 (3) | 3 (4)
Chronic Kidney disease (Renal and urinary disorders) | 2 (5) | 3 (13)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (5) | 2 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (37) | 7 (32)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (4)
Rash acneiform (Skin and subcutaneous tissue disorders) | 3 (7) | 4 (17)
Superficial thrombophlebitis (Vascular disorders) | 2 (3) | 1 (9)
Urinary tract infection (Infections and infestations) | 3 (6) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT02581943/Prot_SAP_000.pdf
  • Informed Consent Form (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT02581943/ICF_001.pdf